CLINICAL TRIAL: NCT04072159
Title: Community Pharmacists Vaccinating Against Cancer (CPVAC): A Pilot Randomized Controlled Trial Aimed at Increasing Human Papillomavirus Vaccine Completion Rates Among Racially/Ethnically Diverse Yout
Brief Title: Community Pharmacists Vaccinate Against Cancer
Acronym: CPVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Adelante Healthcare (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007938; 5U54MD002316-12 (NIH)
Record Dates: First submitted 2019-05-28; First posted 2019-08-28 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Human Papillomavirus Vaccines

STUDY DESIGN:
Intervention Model Description: This pilot intervention is a randomized controlled trial that uses a pre-test/post-test design. Caregivers of HPV vaccine age-eligible minors who are patients of a federally qualified health center, Adelante Healthcare Mesa, will be randomized to Intervention Group (pharmacy), or Control Group (usual care).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-Administered HPV Vaccine Series Completion group (Experimental): For the Pharmacist-Administered HPV Vaccine Series Completion group (intervention group), primary care providers will refer patients who have received the initial HPV vaccine to receive the additional doses at patients' community retail pharmacies. Patients between ages 9-14 will need to receive one additional HPV vaccine dose with their community pharmacist 6-12 months after receiving Dose 1. Patients aged 15 and older will need to receive the 2nd dose 1-2 months after receiving the first HPV vaccine dose and the 3rd dose 6-months after receiving the initial dose.
  Interventions: Behavioral: Community Pharmacists Vaccinating Against Cancer
- Primary Care Provider HPV Vaccine Series Completion (No Intervention): Participant in the Primary Care Provider HPV Vaccine Series Completion (control group) will receive standard care and will be scheduled to return to the clinic for the remaining HPV vaccine doses.

INTERVENTIONS:
Behavioral: Community Pharmacists Vaccinating Against Cancer — Upon completing informed consent, parents of children who have received Dose 1 of the HPV vaccine at the recent clinical visit will be invited to participate in the study. Upon completing the demographic form and pre-test survey for the study, they will be randomized to intervention or control group. Participants in the intervention group will be asked to complete the additional vaccine doses with their community pharmacist. A provider from the participating clinic will electronically prescribe the HPV vaccine dose. Participants in the control group will be scheduled to return to the clinic (based on the vaccine schedule) to complete the vaccine series. The research team will conduct a follow-up survey six months after baseline for each participant. A sample (n=30) of intervention and control group participants will be invited to participate in an in-depth interview to gauge both parents' and children's' acceptability of this intervention.
  Arms: Pharmacist-Administered HPV Vaccine Series Completion group

SUMMARY:
Latino and African American populations have a higher rate of human papillomavirus (HPV) vaccine initiation; however, they have a significantly less likelihood of completing the vaccine series. Pharmacists are licensed to vaccinate against the HPV virus. However, they are less likely to administer the vaccine. Although past research has recommended incorporating pharmacists to increase adolescent vaccination, no intervention studies, to our knowledge, have tested a healthcare delivery model that incorporates pharmacists to complete the HPV vaccine series. The aims of this pilot randomized controlled trial are to 1) determine the preliminary efficacy of an intervention to increase HPV vaccine series completion with the community pharmacist vs. with the primary care provider among racially/ethnically diverse participants, and 2) assess perceived intervention feasibility and acceptability of the intervention among intervention participants and primary care clinic staff.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) is the most common sexually transmitted infection, and persistent infection with oncogenic HPV strains causes cancer. Commercially available 9-valent HPV vaccines offer the potential of immunity against seven oncogenic strains and the two low-risk strains that cause over 90% of genital warts. The majority of HPV-related cancers and genital warts can be prevented through the timely uptake and completion of the HPV vaccine series. However, in 2016 only 37.5% of boys and 49.5% of girls completed the HPV vaccine series, and racial/ethnic minority youth populations are least likely to complete the vaccine series. More specifically, Latino and African American populations have a higher rate of initiation of the vaccine; however, they have a significantly less likelihood of completing the vaccine series. Past research with Latino and African American populations determined the following patient-level barriers to vaccine completion: caregivers' lack of awareness to receive additional vaccine doses, lack of time to attend an additional vaccine-only primary care clinic appointment, and other structural barriers that prohibit caregivers and their children from returning to primary care clinics for additional vaccine doses. Pharmacists are licensed to vaccinate against the HPV virus. However, they are less likely to administer the vaccine. Although past research has recommended incorporating pharmacists to increase adolescent vaccination, no intervention studies, to our knowledge, have tested a healthcare delivery model that incorporates pharmacists to complete the HPV vaccine series. We propose a randomized controlled pilot study titled Community Pharmacists Vaccinate Against Cancer (CPVAC). In CPVAC, the PI will oversample for ethnic minority (particularly African American and Hispanic) HPV vaccine age-eligible children and their caregivers to take part in the study. Patients will be randomized to the Pharmacist-Administered HPV Vaccine Series Completion group or Primary Care Provider HPV Vaccine Series Completion (control) group. After enrolling in the study, primary care providers (PCPs) of patients in the Pharmacist-Administered HPV Vaccine Series Completion group will contact the patients' community pharmacy and prescribe the remaining HPV vaccine dose(s). The pharmacy will electronically update patients' files and schedule the HPV vaccine "refill" (additional doses) at the appropriate dosing schedule. The pharmacy will contact patients' caregivers when it is time to complete additional HPV vaccine dose(s). Primary Care Provider HPV Vaccine Series Completion group participants will receive usual care, returning to their PCPs to complete the additional HPV vaccine doses. The aims of this study are to 1) determine the preliminary efficacy of CPVAC to increase HPV vaccine series completion with the community pharmacist vs. with the primary care provider among racially/ethnically diverse participants, and 2) assess perceived intervention feasibility and acceptability of CPVAC among intervention participants and primary care clinic staff. Findings from this pilot study can be used to inform a larger randomized controlled trial to examine intervention effectiveness and analyze the cost-benefit of working with community pharmacies to enhance HPV vaccine completion among diverse children.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of a child between ages 9-18 who has either not received any HPV vaccine doses or has received only initial HPV dose
* Receives care at Adelante Healthcare Mesa
* Fluent in English and/or Spanish
* Willing to provide informed consent

Exclusion Criteria:

* Caregivers whose child has completed additional HPV vaccine doses
* Child is over age 18 years (no caregiver consent needed)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Adelante Healthcare Mesa, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koskan A, Zittel ME, Lee C, Sanchez O, Alvarez L, Helitzer DL. The feasibility and acceptability of a pilot randomized controlled trial testing pharmacy-based HPV vaccine completion. Res Social Adm Pharm. 2022 Jun;18(6):3038-3045. doi: 10.1016/j.sapharm.2021.08.002. Epub 2021 Aug 8. PMID 34389257

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacist-Administered Human Papillomavirus (HPV) Vaccine Series Completion Group: For the Pharmacist-Administered HPV Vaccine Series Completion group, primary care providers will refer patients who have received the initial HPV vaccine to receive the additional doses at patients' community retail pharmacy. Community Pharmacists Vaccinating Against Cancer: Upon completing informed consent, parents of children who have received Dose 1 of the HPV vaccine at the recent clinical visit will be invited to participate in the study. Upon completing the demographic form and pre-test survey for the study, they will be randomized to intervention or control group. Participants in the intervention group will be asked to complete the additional vaccine doses with their community pharmacist. A provider from the participating clinic will electronically prescribe the HPV vaccine dose. Participants in the control group will be scheduled to return to the clinic (based on the vaccine schedule) to complete the vaccine series. The research team will conduct a follow-up survey six months after baseline for each participant.
- Primary Care Provider HPV Vaccine Series Completion: Primary Care Provider HPV Vaccine Series Completion Group participants will return to the primary care practitioner to complete the HPV vaccine series (usual care).
Period: Overall Study
Arm/Group | Pharmacist-Administered Human Papillomavirus (HPV) Vaccine Series Completion Group | Primary Care Provider HPV Vaccine Series Completion
Started | 16 | 17
Completed | 8 | 11
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pharmacist-Administered HPV Vaccine Series Completion Group: For the Pharmacist-Administered HPV Vaccine Series Completion group, primary care providers will refer patients who have received the initial HPV vaccine to receive the additional doses at patients' community retail pharmacy. Community Pharmacists Vaccinating Against Cancer: Upon completing informed consent, parents of children who have received Dose 1 of the HPV vaccine at the recent clinical visit will be invited to participate in the study. Upon completing the demographic form and pre-test survey for the study, they will be randomized to intervention or control group. Participants in the intervention group will be asked to complete the additional vaccine doses with their community pharmacist. A provider from the participating clinic will electronically prescribe the HPV vaccine dose. Participants in the control group will be scheduled to return to the clinic (based on the vaccine schedule) to complete the vaccine series. The research team will conduct a follow-up survey six months after baseline for each participant.
- Total: Total of all reporting groups
Arm/Group | Pharmacist-Administered HPV Vaccine Series Completion Group | Primary Care Provider HPV Vaccine Series Completion | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Full Range); unit: years] | 37.8 [31 to 53] | 37.1 [30 to 62] | 37.4 [30 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female, Male: Female | 15 | 15 | 30
  Sex: Female, Male: Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 4 | 6
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed HPV Vaccine Series(Preliminary Efficacy)
Description: Whether child completed HPV vaccine series with pharmacist (self-report on post-test and patient medical record)
Time Frame: 6 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-Administered HPV Vaccine Series Completion Group | Primary Care Provider HPV Vaccine Series Completion
Number analyzed (Participants) | 8 | 11
Participants | 8 | 11

2. Secondary Outcome: Intervention Feasibility in Participant Enrollment/Study Completion
Description: Ability to enroll 90 participants into study and retain study participants, ability to retain 90 participants post-intervention (as evidenced by collecting intervention and control group post-tests) - Compare recruitment/enrollment and intervention completion
Time Frame: 1 year after intervention baseline (March 2020)
Measure: Count of Participants; unit: Participants
Groups:
- Pharmacist-Administered HPV Vaccine Series Completion Group: Similar to past HPV vaccine pilot interventions with community pharmacists, our study did not enroll and have a retention rate of sufficient participants to demonstrate feasibility.
Arm/Group | Pharmacist-Administered HPV Vaccine Series Completion Group
Number analyzed (Participants) | 14
Participants | 8

ADVERSE EVENTS:
Time Frame: We monitored adverse events monthly with our study staff when they worked in the clinic from April 2019 - February 2020 (10 months).
Description: We asked clinic staff to report any adverse events related to the study to our study staff. Additionally, in our study informed consent document, we asked participants to notify us (by calling the study principal investigator) of any adverse events.
Arm/Group | Pharmacist-Administered HPV Vaccine Series Completion Group | Primary Care Provider HPV Vaccine Series Completion
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

LIMITATIONS AND CAVEATS:
In the protocol, all parents of HPV vaccine age-eligible children were eligible for recruitment. This changed to only parents of adolescents who vaccinated that day.

Study providers did not recommend the HPV vaccine to children ages 9 and 10. Once the intervention began, clinic providers decided not fax a prescription for additional vaccine doses since pharmacists can administer all vaccine booster doses without a provider prescription.

We ended study recruitment early because of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT04072159/Prot_SAP_000.pdf